CLINICAL TRIAL: NCT01721291
Title: Improving Inhaler Treatment and Small Airways Assessment in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Inhaler Lung Deposition in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIHRCDF; NIHR-CDF-2011-04-053 (Other Grant/Funding Number: UK - NATIONAL INSTITUTE FOR HEALTH RESEARCH); 2011-005544-10 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-11-05 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-05

CONDITIONS: CHRONIC OBSTRUCTIVE PULMONARY DISEASE; ASTHMA; HEALTHY SUBJECTS
Keywords: CHRONIC OBSTRUCTIVE PULMONARY DISEASE; ASTHMA; SALBUTAMOL; ALBUTEROL; VENTOLIN; LUNG PHYSIOLOGY; LUNG DEPOSITION; INHALERS; DRUG THERAPY
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD 1 (Experimental): COPD patients
  Interventions: Drug: SALBUTAMOL
- Healthy (Experimental): Healthy participants
  Interventions: Drug: SALBUTAMOL
- COPD 2 (Experimental): Second group of COPD patients
  Interventions: Drug: SALBUTAMOL
- Asthmatics (Active Comparator): Asthmatics patients
  Interventions: Drug: SALBUTAMOL

INTERVENTIONS:
Drug: SALBUTAMOL — In the LUNG DEPOSITION STUDY; SALBUTAMOL INHALED VIA RESEARCH NEBULISER at 3 PARTICLES SIZES OF 1.5 MICRONS, 3 MICRONS AND 6 MICRONS WILL BE GIVEN AT SLOW INHLATION AND AGAIN AT FAST INHALTION;DOSAGE- 30 MICROGRAMS, ONE SINGLE INHALATION ONLY. IN ADDITION, SALBUTAMOL AT 200 MICROGRAMS INHALED VIA A STANDARD METERED DOSE INHALER WILL ALSO BE GIVEN AS A SINGLE INHALATION.
  In the LUNG PHYSIOLOGY STUDY; SALBUTAMOL INHALED VIA RESEARCH NEBULISER at 3 PARTICLES SIZES OF 1.5 MICRONS, 3 MICRONS AND 6 MICRONS WILL BE GIVEN AT TWO DOSAGES OF 30 MICROGRAMS AND AGAIN AT 15 MICROGRAMS, ONE SINGLE INHALATION ONLY. IN ADDITION, SALBUTAMOL AT 200 MICROGRAMS INHALED VIA A STANDARD METERED DOSE INHALER WILL ALSO BE GIVEN AS A SINGLE INHALATION. ALL INHALATIONS WIL BE AT SLOW INHALTION IN THIS PART OF THE STUDY.
  Other Names: ALBUTEROL; VENTOLIN; SALMOL

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) experience breathing difficulties because the airways deep in their lungs become narrowed. COPD patients use inhaler drugs to provide relief from breathlessness. However, current inhalers are inefficient as they deliver a 'coarse-mist' of drug-droplets that do not reach the deep airways.

In our study, we will use an inhaler of 'fine-mist' drug-droplets, tagged with a radioactive tracer to track them. We will take images of the lungs to see if the fine-mist droplets reach the deep airways, and assess if this improves the breathing capacity in our patients. Our research may allow the development of new, more efficient inhalers to improve treatment for patients with COPD.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of the research (or "knowledge gap" this research is designed to fill) is to understand the fate of inhaled drug within the lungs of COPD patients. Current inhalers in use were developed to treat asthma, which is predominantly a disease of the large airways, and these inhalers may not be optimal in treating COPD patients (which is predominantly a disease of the small airways). Poor delivery of inhaled bronchodilators to the peripheral deep airways may be a major factor limiting the clinical benefit provided by existing devices. The key to successful treatment could be to accurately target inhaled drug to the diseased lung sites, which is the hypothesis that this protocol will test.

DESIGN & FUNDING:

Dr Omar Usmani has developed the research protocol and the study has been funded by the UK Government Department of Health through the NIHR (National Institute for Health Research), which funds leading edge research in the NHS focussed on the needs of patients and the public and aims to improve the health and wealth of the nation through research. The study has been peer reviewed by International Experts in this field of research.

PROTOCOL:

This protocol has two studies: Lung DEPOSITION study (in COPD patients and Healthy subjects) and Lung PHYSIOLOGY study (in COPD patients and Asthmatics).

Each study (Lung DEPOSITION and Lung PHYSIOLOGY) will be a randomised, double-blind, crossover, (7 treatments,controlled against pMDI salbutamol), study. Treatments will be given as one off dose administration.

There will be an interval of at least 5 days between each study visit. The Lung DEPOSITION study will involve radiolabelled drug treatments.

All the treatments in the LUNG PHYSIOLOGY study will be non-radiolabelled. Salbutamol will be the drug aerosol administered to each subject at each visit. Subjects and investigators will be blinded to the 'fine-mist' aerosol particle sizes given (at 6 treatments). The control arm will be salbutamol drug aerosol delivered as a 'coarse mist' standard metered dose inhaler (7th treatment visit).

RECRUITMENT/SAMPLE SIZE; The study will recruit; Lung DEPOSITION study: 12 mild-moderate COPD patients, 12 healthy subjects Lung PHYSIOLOGY study: 26 mild-moderate COPD patients, 13 mild-moderate asthmatic patients

INCLUSION / EXCLUSION:

At the screening vist, no one will be unfairly excluded from the research, particularly as COPD is a disease of older age and those over 65 should not be discriminated against. This research will therefore reflect the 'real world' of COPD.

ELIGIBILITY:
Inclusion Criteria:

- COPD patients, either male or female, over the age of 40 with a clinical diagnosis of COPD with airflow obstruction(FEV1/FVC<0.7) and post-bronchodilator FEV1>50% predicted, gas trapping (on lung volume testing), and decreased carbon monoxide transfer factor.

Healthy subjects will be nonsmokers(or exsmokers stopped 5 years ago), will have no respiratory disease, normal spirometry and be age-matched to the COPD patients.

Asthmatic subjects, either male or female, over the age of 18 with a clinical diagnosis of Asthma with airflow obstruction (FEV1/FVC<0.7).

All patients should be capable of giving informed consent.

Exclusion Criteria:

1. Oral corticosteroids taken within last month.
2. Current involvement (or involvement in the last 4 weeks)in clinical trials assessing investigational medicinal products.
3. Previous adverse reaction to short or long acting β2 agonist.
4. Any subject with a contraindication to taking inhaled beta2-adrenoceptor agonists (especially salbutamol) as listed in the British National Formulary will not be entered into this study.
5. Those who have experienced an acute respiratory exacerbation requiring emergency room treatment and/ or hospitalisation within four weeks of visit 1 (screening visit).
6. Pregnant or breastfeeding women.
7. Subjects unable to give Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar S USMANI, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital & Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Usmani OS, Biddiscombe MF, Barnes PJ. Regional lung deposition and bronchodilator response as a function of beta2-agonist particle size. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1497-504. doi: 10.1164/rccm.200410-1414OC. Epub 2005 Sep 28. PMID 16192448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This protocol has two studies: Lung DEPOSITION study (in COPD patients and Healthy subjects) and Lung PHYSIOLOGY study (in COPD patients and Asthmatics).
Groups:
- COPD- Lung DEPOSITION Study: Lung DEPOSITION study COPD patients All participant received SALBUTAMOL INHALED VIA RESEARCH NEBULISER at 3 PARTICLES SIZES OF 1.5 MICRONS, 3 MICRONS AND 6 MICRONS GIVEN AT SLOW INHLATION AND AGAIN AT FAST INHALTION;DOSAGE- 30 MICROGRAMS, ONE SINGLE INHALATION ONLY. IN ADDITION, SALBUTAMOL AT 200 MICROGRAMS INHALED VIA A STANDARD METERED DOSE INHALER GIVEN AS A SINGLE INHALATION.
- Healthy - Lung DEPOSITION Study: Lung DEPOSITION study
  Healthy participants received:
  SALBUTAMOL INHALED VIA RESEARCH NEBULISER at 3 PARTICLES SIZES OF 1.5 MICRONS, 3 MICRONS AND 6 MICRONS GIVEN AT SLOW INHLATION AND AGAIN AT FAST INHALTION;DOSAGE- 30 MICROGRAMS, ONE SINGLE INHALATION ONLY. IN ADDITION, SALBUTAMOL AT 200 MICROGRAMS INHALED VIA A STANDARD METERED DOSE INHALER GIVEN AS A SINGLE INHALATION.
Period: Overall Study
Arm/Group | COPD- Lung DEPOSITION Study | Healthy - Lung DEPOSITION Study
Started | 14 | 12
Completed | 12 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — did not like the treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- COPD: COPD patients
- Total: Total of all reporting groups
Arm/Group | COPD | Healthy | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Full Range); unit: years] | 66.08 [56 to 77] | 64.08 [50 to 76] | 65.08 [50 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 12 | 65
Force experation in 1s (FEV1) [Mean (Full Range); unit: litre] | 1.63 [0.97 to 2.24] | 2.55 [1.55 to 3.76] | 2.12 [0.71 to 3.9]

OUTCOME MEASURES:

1. Primary Outcome: ANALYSIS OF LUNG DEPOSITION - Penetration Index
Description: Images of the lungs will be taken for radiolabelled salbutamol treatment. The images will be processed using computer software and the lungs divided into central airways (C - region) and peripheral airways (P -region). We will analyse the amount of radiolabelled salbutamol in each region and calculate how deep into the lungs the inhaled salbutamol has reached by using the ratio C/P which is known as the Penetration Index.
Time Frame: 5 MINUTES AFTER INHALATION OF SALBUTAMOL
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Healthy_1.5um Slow: Healthy participants Salbutamol 1.5um slow
- Healthy_1.5um Fast: Healthy participants Salbutamol 1.5um fast
- COPD 1_1.5um Slow: COPD patients Salbutamol 1.5um slow
- COPD1_1.5um Fast: Second group of COPD patients Salbutamol 1.5um fast
- Healthy_3um Slow: Healthy participants Salbutamol 3um slow
- Healthy_3um Fast: Healthy participants Salbutamol 3um fast
- COPD_3um Slow: COPD patients Salbutamol 3um slow
- COPD_3um Fast: COPD patients Salbutamol 3um fast
- Healthy_6um Slow: Healthy participants Salbutamol 6um slow
- Healthy_6um Fast: Healthy participants Salbutamol 6um fast
- COPD_6um Slow: COPD patients Salbutamol 6um slow
- COPD_6um Fast: COPD patients Salbutamol 6um fast
Arm/Group | Healthy_1.5um Slow | Healthy_1.5um Fast | COPD 1_1.5um Slow | COPD1_1.5um Fast | Healthy_3um Slow | Healthy_3um Fast | COPD_3um Slow | COPD_3um Fast | Healthy_6um Slow | Healthy_6um Fast | COPD_6um Slow | COPD_6um Fast
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
ratio | 0.8 (0.08) | 0.72 (0.12) | 0.69 (0.13) | 0.58 (0.14) | 0.75 (0.11) | 0.63 (0.15) | 0.65 (0.18) | 0.48 (0.16) | 0.51 (0.1) | 0.46 (0.04) | 0.37 (0.12) | 0.32 (0.08)

ADVERSE EVENTS:
Time Frame: 6 month
Groups:
- Healthy_1.5um Slow: Healthy participants received Salbutamol 1.5um slow - Lung DEPOSITION study
- Healthy_1.5um Fast: Healthy participants received Salbutamol 1.5um fast - Lung DEPOSITION study
- COPD_1.5um Slow: Participants with COPD received Salbutamol 1.5um slow - Lung DEPOSITION study
- COPD_1.5um Fast: Participants with COPD received Salbutamol 1.5um fast - Lung DEPOSITION study
- Healthy_3um Slow: Healthy participants received Salbutamol 3um slow - Lung DEPOSITION study
- Healthy_3um Fast: Healthy participants received Salbutamol 3um fast - Lung DEPOSITION study
- COPD_3um Slow: Participants with received COPD Salbutamol 3um slow - Lung DEPOSITION study
- COPD_3um Fast: Participants with COPD Salbutamol 3um fast - Lung DEPOSITION study
- Healthy_6um Slow: Healthy participants received Salbutamol 6um slow - Lung DEPOSITION study
- Healthy_6um Fast: Healthy participants received Salbutamol 6um fast - Lung DEPOSITION study
- COPD_6um Slow: Participants with COPD received Salbutamol 6um slow - Lung DEPOSITION study
- COPD_6um Fast: Participants with COPD received Salbutamol 6um fast - Lung DEPOSITION study
Arm/Group | Healthy_1.5um Slow | Healthy_1.5um Fast | COPD_1.5um Slow | COPD_1.5um Fast | Healthy_3um Slow | Healthy_3um Fast | COPD_3um Slow | COPD_3um Fast | Healthy_6um Slow | Healthy_6um Fast | COPD_6um Slow | COPD_6um Fast
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/14 | 0/14 | 0/12 | 0/12 | 0/14 | 0/14 | 0/12 | 0/12 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/14 | 0/14 | 0/12 | 0/12 | 0/14 | 0/14 | 0/12 | 0/12 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/14 | 1/14 | 0/12 | 0/12 | 1/14 | 0/14 | 1/12 | 0/12 | 1/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy_1.5um Slow (N=12) | Healthy_1.5um Fast (N=12) | COPD_1.5um Slow (N=14) | COPD_1.5um Fast (N=14) | Healthy_3um Slow (N=12) | Healthy_3um Fast (N=12) | COPD_3um Slow (N=14) | COPD_3um Fast (N=14) | Healthy_6um Slow (N=12) | Healthy_6um Fast (N=12) | COPD_6um Slow (N=14) | COPD_6um Fast (N=14)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoe (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulled muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operatoin (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT01721291/Prot_SAP_000.pdf